CLINICAL TRIAL: NCT02016664
Title: Plasma Concentration of Ketamine and Norketamine in Patients on Oral Ketamine for Chronic Neuropathic Pain : A Pilot Study.
Brief Title: Plasma Concentration of Ketamine and Norketamine .
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Qutaiba Tawfic, Clinical Fellow, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: OKPCS
Record Dates: First submitted 2013-12-16; First posted 2013-12-20 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Chronic Pain
Keywords: Chronic Pain, Ketamine, Safety
MeSH Terms: conditions — Chronic Pain | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chronic pain patients on oral ketamine (Experimental): Days 1-7:
  Subjects will be given a 7 day supply of 10 mg ketamine tablets three times per day for seven days and to return to clinic on Day 7. They will be instructed not to take their morning dose of ketamine and to eat a light breakfast on Day 7. Upon arrival, the patient will have a 20 gauge (saline locked) IV started in the antecubital fossa to allow for five blood samples: Time Zero,30, 60,90 and 120 minutes. The first blood sample at Time 0 will be obtained just before the patient takes his/her oral dose of ketamine.
  Days 8-14:
  The subjects will be given a supply of 20 mg ketamine capsules and instructed to take them three times per day, at specified times, and to return to clinic on Day 14. The instructions and procedures at the second clinic visit will be the same as on Day 7.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — The St.Joseph's Heath Care Pharmacy will supply the compounded oral ketamine capsules. Patients who are going to participate in this study are already taking this oral ketamine as a part of their chronic pain medications. No new patient will start oral ketamine for the sake of this study. Two doses of oral ketamine will be used for the same patient, 10 mg and 20 mg every 8 hours. These doses are the standard doses in our clinic. Other clinics using much higher doses.

SUMMARY:
Oral ketamine is increasingly used by doctors to both reduce the amount of narcotic pain medication consumed and to improve chronic pain management in difficult cases. How much is absorbed when taken orally, as opposed to intravenously ,is unknown. Ketamine may cause sedation, and occasionally cognitive impairment. Therefore, there are safety concerns associated with its usage as an out-patient may engage in activities where cognitive impairment is dangerous,such as driving. This study is designed to measure the plasma concentrations of ketamine and its active metabolite, norketamine, in people taking low dose oral ketamine for chronic pain. The goal of the study is to verify that low dose oral ketamine produces plasma concentrations below the level associated with toxic symptoms,and thus can be safely used long-term for the treatment of chronic pain .

DETAILED DESCRIPTION:
This is a non-randomized, cohort study to measure the serum uptake of low dose oral ketamine in chronic pain patients. The SJHC pharmacy has a list of patients to whom they dispense oral ketamine. We plan to recruit fifteen patients from this patient group.

This is a pilot study and very little information is available to help with sample size calculations. We also plan to measure change in mean pain score from Day to Day 14 using the Brief Pain Inventory (BPI) This data will aid the design and calculation of sample size in future studies. Study Design: Days 1-7: Following informed consent, the patient's demographic information and initial assessment will be completed on Day 1 at the first visit. They will be allowed to continue all usual systemic analgesic medications. They will be given instructions on how to take the study medication and will be given a list of foods that could possibly induce or inhibit the enzyme, Cyp3A4 or Cyp2B6 (i.e. grapefruit or grapefruit juice). Subjects will be given a 7 day supply of 10 mg ketamine tablets. The patients will be instructed to take one ketamine tablet three times per day at specified times for seven days and to return to clinic on Day 7. They will be instructed not to take their morning dose of ketamine and to eat a light breakfast on Day 7. Upon arrival, the patients will complete the Brief Pain Inventory and side effects questionnaire. The patient will have a 20 gauge (saline locked) IV started in the antecubital fossa to allow for five blood samples: Time Zero, 30, 60, 90 and 120 minutes. The first blood sample at Time 0 will be obtained just before the patient takes his/her oral dose of ketamine (trough concentration). The four remaining samples will be taken after the patient ingests his/her 10 mg ketamine dose. Time Activity Arrival Complete BPI, side effect questionnaire Time Zero Blood draw, then take 10mg oral ketamine dose 30 minutes post ingestion Blood draw 60 minutes post ingestion Blood draw 90 minutes post ingestion Blood draw 120 minutes post-ingestion Blood Draw Days 8-14: The subjects will be given a supply of 20 mg ketamine capsules and instructed to take them three times per day, at specified times, and to return to clinic on Day 14. The instructions and procedures at the second clinic visit will be the same as on Day 7.

ELIGIBILITY:
Inclusion Criteria:

* Patient currently takes oral ketamine for the treatment of chronic neuropathic pain.
* Age >18 and < 75 years
* Both males and females 4.Ability to speak English adequately to understand the consent and participate in the study
* No other route of ketamine within past 7 days (Topical/IV)

Exclusion Criteria:

* Patient receiving liver enzyme inducers or inhibitors of Cytochrome CYP3A4, or CYP2B6 like clarithromycin, rifampin, and recent ingestion of grapefruit juice.
* Patients who have had gastric bypass surgery
* Patients who did not follow the prescribed protocol
* Renal Failure defined as Creatinine Clearance <50 mL/min
* Hepatic insufficiency by history

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Plasma level of oral ketamine and norketamine at two different doses. | 0,30,60,90 and 120 min after ingestion.
  Plasma level of ketamine and norketamine will be tested just before ingestion of oral ketamine (trough level) and then after at 30,60,90 and 120min. Patients will be already using oral ketamine therapy for 7 days before the test. This test will be repeated twice on 2 different doses (10 and 2o mg q 8 hr).

SECONDARY OUTCOMES:
Mean Pain Score | week 1 and week 2
  Mean pain score will be recorded at the end of one week of ingestion for each dose.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Morley-Foster, MD, FRCPC, Principal Investigator — Department of Anesthesia and Perioperative Medicine, Western University, Canada.
Locations (1):
- St.Joseph's Health Care, Western University, London, Ontario, Canada